CLINICAL TRIAL: NCT06807463
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2a Trial to Characterize the Efficacy and Safety of TEV-53408 in Adults With Celiac Disease While Undergoing Oral Gluten Exposure
Brief Title: A Trial to Assess the Efficacy and Safety of TEV-53408 in Adults With Celiac Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV53408-IMM-20042; 2024-517081-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEV-53408 (Experimental)
  Interventions: Drug: TEV-53408
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-53408 — Solution for subcutaneous (sc) injection
  Arms: TEV-53408
Drug: Placebo — Solution for subcutaneous (sc) injection
  Arms: Placebo

SUMMARY:
The primary efficacy objective of the trial is to assess the ability of TEV-53408 to attenuate gluten-induced enteropathy in adults with celiac disease.

The primary safety objective of the trial is to assess the safety of TEV-53408 in adults with celiac disease.

A secondary objective is to further assess the efficacy of TEV-53408 in adults with celiac disease.

The expected trial duration per participant is approximately 86 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease at least 12 months prior to screening
* On a gluten-free diet for at least 12 months prior to screening
* Women must not be pregnant, lactating, breastfeeding, or planning pregnancy during the trial period
* Male participants (including vasectomized) with women of child-bearing potential partners (whether pregnant or not) must use condoms and also agree not to donate sperm for the designated period

NOTE - Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* A diagnosis or suspicion of refractory celiac disease
* History of severe celiac-related symptoms following gluten exposure that require acute medical care or intervention of a health care professional
* Any other gastrointestinal disease or condition that may interfere with the assessment of celiac disease
* Current or history of malignancy or treatment of malignancy in the last 5 years, excluding treated basal cell carcinoma
* Pregnant or lactating woman, or plans to become pregnant during the trial; any man who is considering fathering a child or donating sperm during the trial
* A history of chronic alcohol or substance abuse disorder within the previous 2 years.
* An active infection(s) requiring treatment with intravenous (iv) anti-infectives (antibiotics, antivirals, antifungals) within 30 days prior to screening or oral anti-infectives (antibiotics, antivirals, antifungals) within 14 days prior to screening
* Received or intends to receive any live vaccine within 4 weeks or any non-live vaccine 2 weeks prior to investigational medicinal product administration.

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Villous Atrophy as Measured by Villous Height to Crypt Depth Ratio (Vh:Cd) | Baseline, Week 8
  Vh:Cd is used to assess the severity of celiac disease. It is calculated by dividing the villous height by the crypt depth. A lower ratio indicates more damage.
Number of Participants With at Least One Treatment-Emergent Adverse Event | Up to Week 28
Number of Participants With at Least One Treatment-Emergent Serious Adverse Event | Up to Week 28
Number of Participants With at Least One Protocol-Defined Adverse Event of Special Interest (PDAESI) | Up to Week 28
Number of Participants Who Discontinued From the Study Due to an Adverse Event | Up to Week 28

SECONDARY OUTCOMES:
Change From Baseline in Intraepithelial Lymphocyte (IEL) Density | Baseline, Week 8
Change From Baseline in the VCIEL score | Baseline, Week 8
  VCIEL score is a calculation using the standardized Vh:Cd and standardized IEL. The standardized Vh:Cd is calculated as the difference between the mean Vh:Cd subtracted from each Vh:Cd divided by the Vh:Cd standard deviation. The standardized IEL is calculated as the difference between the mean IEL subtracted from each IEL divided by the IEL standard deviation. VCIEL is the standardized Vh:Cd minus the standardized IEL.

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (21):
- United States (16):
  - Teva Investigational Site 12138, Murrieta, California
  - Teva Investigational Site 12131, Colorado Springs, Colorado
  - Teva Investigational Site 12134, Inverness, Florida
  - Teva Investigational Site 12126, Miami Lakes, Florida
  - Teva Investigational Site 12135, New Port Richey, Florida
  - Teva Investigational Site 12130, Atlanta, Georgia
  - Teva Investigational Site 12133, Marrero, Louisiana
  - Teva Investigational Site 12132, Clinton Township, Michigan
  - Teva Investigational Site 12121, Wyoming, Michigan
  - Teva Investigational Site 12129, Rochester, Minnesota
  - Teva Investigational Site 12128, New York, New York
  - Teva Investigational Site 12125, Greenville, North Carolina
  - Teva Investigational Site 12127, Winston-Salem, North Carolina
  - Teva Investigational Site 12137, Waco, Texas
  - Teva Investigational Site 12122, Ogden, Utah
  - Teva Investigational Site 12123, Lynchburg, Virginia
- Australia (3):
  - Teva Investigational Site 78139, Fitzroy
  - Teva Investigational Site 78140, Maroochydore
  - Teva Investigational Site 78137, Midland
- Finland (2):
  - Teva Investigational Site 40063, Helsinki
  - Teva Investigational Site 40062, Tampere

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.